CLINICAL TRIAL: NCT06845605
Title: A Qualitative Exploration Study of Healthcare Professionals' Perspectives in Haemodialysis Needling to Enhance Patients' Overall Experience
Brief Title: Behind the Needle: Healthcare Professionals' Perspectives on HD Needling
Status: Recruiting | Type: Observational
Sponsor: East and North Hertfordshire NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: RD2024-55
Record Dates: First submitted 2024-10-30; First posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2024-10

CONDITIONS: Perspective of Healthcare Professionals Haemodialysis Needling; Dialysis
Keywords: Haemodialysis; Haemodialysis needling; End-Stage Renal Disease; Fistula; Cannulation
MeSH Terms: conditions — Kidney Failure, Chronic; Fistula

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Haemodialysis is essential for patients with End-Stage Renal Disease (ESRD), requiring consistent vascular access through arteriovenous fistulas or grafts. This involves frequent needling, a procedure that is painful and distressing for many patients, causing significant emotional and physical demands on healthcare professionals working in the dialysis units. In the UK, about 30,000 patients receive haemodialysis, involving over 300 needling procedures annually.

Healthcare professionals (Registered nurses and healthcare assistants) play a crucial role, with their expertise directly affecting patient outcomes. However, 60% of HCPs (healthcare professionals) report high job-related stress, particularly due to needling demands. Effective needling requires not only technical proficiency but also managing patient pain and anxiety. Strong staff-patient relationships, characterized by empathy and understanding, can enhance the needling experience. Challenges for dialysis unit staff includes the technical difficulty of needling and the emotional burden of patient care. Studies highlight the need for better training and support systems to help them cope with these demands.

Understanding healthcare professionals' perspectives can identify areas for improvement, inform training programs, and improve experiences in dialysis units. Research by Rahmah et al. (2018) and Duncanson (2023) emphasizes the importance of HCPs skills and the psychological toll on them, suggesting further exploration of this area is needed. The primary aim of this research is to examine HCPs perspectives on the needling experience in haemodialysis, aiming to identify improvement areas and inform targeted training programs to enhance patient experiences. The study will utilize a qualitative exploratory design with semi-structured interviews to gather in-depth insights from HCPs. Data will be collected from renal dialysis units at East and North Hertfordshire NHS Trust, involving 12 to 16 registered nurses performing needling procedures. Thematic analysis will be used to analyse interview transcripts and identify key themes related to technical skills, communication barriers, and patient-related factors. The study will run for 10 months.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be registered nurses or Band 3 healthcare assistants who perform needling procedures in a haemodialysis unit.
* Participants must be employed at the renal dialysis units of East and North Hertfordshire NHS Trust (ENHT), including both the main unit and its satellite units.
* Participants must be willing to participate in the study and share their experiences.
* Participants must be able to speak English fluently to ensure they can communicate effectively, providing rich and comprehensive information.

Exclusion Criteria:

•Registered nurses or healthcare assistants who do not perform needling procedures in a haemodialysis unit will not be eligible to participate.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All data will be collected in the renal dialysis units of ENHT consisting of one main unit and four satellite units. The service provides in-centre haemodialysis to over 600 patients. Eligible nursing staff will be drawn from all service dialysis units.
  The study aims to recruit between 12 to 16 HCPs (registered nurses and healthcare assistants) from dialysis units within East and North Hertfordshire NHS Trust (ENHT). The sample size will be determined based on the concept of information power, ensuring that the data collected is sufficient to address the research questions effectively.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Estimated)
Dates: Start 2024-10-30 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Healthcare professionals' (registered nurses and healthcare assistants) perspectives on the needling experience, with a focus on identifying areas for improvement and informing targeted training programs to enhance the overall patient experience. | March 2024

CONTACTS AND LOCATIONS:
Locations (1):
- East and North Hertfordshire NHS Trust, Stevenage, Hertfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sutton J, Austin Z. Qualitative Research: Data Collection, Analysis, and Management. Can J Hosp Pharm. 2015 May-Jun;68(3):226-31. doi: 10.4212/cjhp.v68i3.1456. No abstract available. PMID 26157184
- [Background] Manoochehri H, Imani E, Atashzadeh-Shoorideh F, Alavi-Majd A. Competence of novice nurses: role of clinical work during studying. J Med Life. 2015;8(Spec Iss 4):32-38. PMID 28316703
- [Background] Hagerty TA, Samuels W, Norcini-Pala A, Gigliotti E. Peplau's Theory of Interpersonal Relations: An Alternate Factor Structure for Patient Experience Data? Nurs Sci Q. 2017 Apr;30(2):160-167. doi: 10.1177/0894318417693286. PMID 28899257
- [Background] Duncanson EL, Chur-Hansen A, Le Leu RK, Macauley L, Burke ALJ, Donnelly FF, Collins KL, McDonald SP, Jesudason S. Dialysis Needle-Related Distress: Patient Perspectives on Identification, Prevention, and Management. Kidney Int Rep. 2023 Sep 14;8(12):2625-2634. doi: 10.1016/j.ekir.2023.09.011. eCollection 2023 Dec. PMID 38106606
- [Background] Rahmah NM, Hariyati TS, Sahar J. Nurses' efforts to maintain competence: a qualitative study. J Public Health Res. 2021 Dec 1;11(2):2736. doi: 10.4081/jphr.2021.2736. PMID 35244357
- [Background] Napalkov P, Felici DM, Chu LK, Jacobs JR, Begelman SM. Incidence of catheter-related complications in patients with central venous or hemodialysis catheters: a health care claims database analysis. BMC Cardiovasc Disord. 2013 Oct 16;13:86. doi: 10.1186/1471-2261-13-86. PMID 24131509
- [Background] Alsbrooks K, Hoerauf K. Prevalence, causes, impacts, and management of needle phobia: An international survey of a general adult population. PLoS One. 2022 Nov 21;17(11):e0276814. doi: 10.1371/journal.pone.0276814. eCollection 2022. PMID 36409734
- [Background] Hill K, Sharp R, Childs J, Esterman A, Le Leu R, Juneja R, Jesudason S. Cannulation practices at haemodialysis initiation via an arteriovenous fistula or arteriovenous graft. J Vasc Access. 2020 Sep;21(5):573-581. doi: 10.1177/1129729819869093. Epub 2019 Aug 18. PMID 31423945
- [Background] Lamb PC, Norton C. Nurses experiences of using clinical competencies a qualitative study. Nurse Educ Pract. 2018 Jul;31:177-181. doi: 10.1016/j.nepr.2018.06.006. Epub 2018 Jun 12. PMID 29929090
- [Background] Fielding C, Bramley L, Stalker C, Brand S, Toft S, Buchanan H. Patients' experiences of cannulation of arteriovenous access for haemodialysis: A qualitative systematic review. J Vasc Access. 2023 Sep;24(5):1121-1133. doi: 10.1177/11297298211067630. Epub 2022 Jan 16. PMID 35034481
- [Background] Bello AK, Okpechi IG, Osman MA, Cho Y, Htay H, Jha V, Wainstein M, Johnson DW. Epidemiology of haemodialysis outcomes. Nat Rev Nephrol. 2022 Jun;18(6):378-395. doi: 10.1038/s41581-022-00542-7. Epub 2022 Feb 22. PMID 35194215
- See also: Moore, C., Ellis-Caird, H., Fielding, C., et al. (2024). Patients' perspectives on key aspects influencing needling for haemodialysis: A qualitative study. Manuscript in preparation — https://salford.figshare.com/collections/_/7366282
- See also: Edgar, Denise & Wilson, Valerie & Moroney, Tracey. (2020). Which is it, person-centred culture, practice or care? It matters. International Practice Development Journal, 10, 1-17. 10.19043/ipdj.101.008. — https://www.fons.org/wp-content/uploads/2024/02/IPDJ_10_01_08.pdf
- See also: Braun V, Clarke V. Using thematic analysis in psychology. Qualitative Research in Psychology. 2006;3(2):77-101 — https://www.researchgate.net/publication/235356393_Using_thematic_analysis_in_psychology